CLINICAL TRIAL: NCT03746626
Title: What Difference do Chaplains Make: Analysis of Chaplain Interventions in Palliative Care in United Kingdom
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Edinburgh Napier University (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Austyn Snowden, Professor in Mental Health, Edinburgh Napier University
Other Study IDs: SHSC 18001
Record Dates: First submitted 2018-11-13; First posted 2018-11-20 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Spirituality; Palliative Care
Keywords: Spiritual care; Palliative care; Chaplain; Day care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Hospice 1: Strathcarron Hospice, Scotland. All consenting patients will either see chaplain or not as many times as per their choice, over eight week stay in day care at the hospice.
  Interventions: Behavioral: Chaplain visit
- Hospice 2: Arthur Rank Hospice, England. All consenting patients will either see chaplain or not as many times as per their choice, over eight week stay in day care at the hospice.
  Interventions: Behavioral: Chaplain visit
- Hospice 3: All consenting patients will either see chaplain or not as many times as per their choice, over eight week stay in day care at the hospice.
  Interventions: Behavioral: Chaplain visit

INTERVENTIONS:
Behavioral: Chaplain visit — The patients will all see a chaplain routinely during 8-week stay according to their personal preference. The chaplain records the 'depth' and frequency of these encounters.

SUMMARY:
Naturalistic pre-post survey design. People with palliative care needs referred to day care in participating hospices will be invited to participate in the study. Those consenting to take part will complete a baseline survey consisting of demographic data on age, gender, reason for admission and whether they self report as religious, spiritual, both, or neither. They also complete he Scottish Patient Reported Outcome Measure (PROM), a five item measure of spiritual outcome/well-being and a free text box. The patient then attends the day care for eight weeks, during which time they may see a chaplain regularly, infrequently, or not at all, entirely dependent on personal preference. The study is designed to be as naturalistic as possible. At the end of the 8 weeks patients complete a follow-up survey containing the same surveys as previous, plus four items about their experiences (or not) with the chaplain. During these eight weeks the chaplain also records the frequency and their interpretation of the depth of the visits with the patient. The primary purpose of the study is to explore the relationship between any change in Scottish PROM scores and the a) frequency and b) chaplain reported depth of the encounters. Secondary objectives are to examine the relationship between the change in PROM scores and the patient's experience of the chaplain interventions. It is hypothesised that the better the chaplain and/or patient self reported experience of the chaplain the greater the improvement in PROM scores. Whether there is any relationship between improvement in PROM scores and whether the patient self describes as religious, spiritual, both or neither will also be analysed.

DETAILED DESCRIPTION:
BACKGROUND: Day-care and Chaplains Hospice day-care can be for patients who have a palliative diagnosis and would benefit from multidisciplinary team (MDT) input, but don't require in patient care. The chaplain's role is to support patients with any spiritual issues they may have. For a number of patients this may be a time for them to begin to understand the limitations that their condition may place upon them, and those may be the issues that they are wanting to explore, along with the implications for them and their families for the future. Some may not want to see a chaplain at all, of course. Faith and religion may play a part here.

There is evidence that patients who talk to chaplains benefit in a number of ways. A recent study showed that being with a chaplain was associated with patients feeling they had a more positive outlook, were less anxious and felt more in control. Anecdotal feedback from General Practitioners (GP)s suggested that that chaplains prevented them prescribing anxiolytics in some cases, reduced unnecessary onward referrals and reduced attendance at surgery. However, it remains unknown what sort of person benefits most from chaplaincy. Further, it is not known whether more or less chaplaincy is better. Likewise, the depth of the connection between patient and chaplain would surely have an impact on the outcome. This study is designed to explore these issues systematically.

Aim

To evaluate the impact of chaplains on patient reported outcomes in palliative day care.

Primary objective:

1. Articulate the a) quantitative and b) qualitative difference chaplains make on patient outcomes.

   Secondary objectives:
2. Understand the relationship between the personal experience of the chaplain encounter(s) and their outcome.
3. Explore the relationship between self-reported spirituality/religion and outcome.

Hypotheses

Primary hypotheses:

1. There will be a significant correlation between the number of times a chaplain sees a patient and the change in PROM scores from baseline to post intervention.
2. There will be a significant correlation between the chaplain reported depth of the encounters and the change in PROM scores from baseline to post intervention.

Secondary hypotheses:

1. The patient experience of the chaplain encounter will be associated with the outcome of that intervention.
2. There will be no difference in Scottish PROM scores according to whether patients self-describe as religious, spiritual, both, or neither.

METHOD: Measures

The Scottish PROM The Scottish PROM is a five-item measure of the outcomes of spiritual care as delivered by a chaplain. It has Likert responses to items concerning how the patient has been in the last two weeks in relation to: peace, control, outlook, anxiety and honesty. It also contains a free text box for elaboration.

Health Related Quality of Life (EQ5D-3L) A short, well validated measure of patient reported health related quality of life. This will be used to explore the impact the patient's health related quality of life has on any findings.

The patient's experience of the chaplain Measuring the experience of the chaplain encounter involves four Likert style question focusing on the chaplain's capacity to facilitate: listening, being able to talk about what is on my mind, understanding and having my faith/beliefs valued.

The chaplain's experience of the encounter The chaplain completes the same questionnaire as the patient, as if they were the patient. They also estimate the 'depth' of the encounter on a 1 to 5 scale devised by a local hospice, with one representing the briefest of encounter to five representing support and prayer at death, to both patient and relatives.

METHOD: Participants

Chaplains Chaplains will be accredited members with national association or equivalent. Volunteers or non-professional chaplains will not be included as 'chaplains' in this study.

Project participants will be patients who have attended the hospices as day patients. Generally speaking all of these hospices support people who are aged 18 years and above living with a life-limiting illness and those who will need end-of-life care. This includes a wide range of conditions from cancer to degenerative neurological conditions to even heart failure. Age ranges are from 18 although in most instances the majority of patients will be above 40 years of age with the number increasing for each decade with the largest group commonly being the 70-80 age group. Most day patients are referred to the hospice through GPs.

Inclusion/exclusion criteria Everybody as described above with the exception of children under 18 or people unable to consent. People who cannot speak English will be supported to participate by relatives or other translator wherever possible.

METHOD: PROCESS First, all patients attending day care for the first time are given a short introductory leaflet, to let them know a study is going on at the hospice, and their participation would be welcome. They take this leaflet home with them. The following week, (week 2), the study 'champion' asks the patient if they would be willing to take part in the study. If the person agrees, they are next asked to read the patient information sheet, complete the consent form and the Baseline questionnaire.

The intervention The chaplain is the intervention. He/she operates as usual, seeing people spontaneously or as they normally would. This is so the study can analyse the impact of chaplaincy as naturally as possible.

The role of the champion is to make sure that the chaplain makes a record of the visits they have had in any given day, paying particular attention to the 'depth' of the interventions. These should be recorded regularly, at the end of every day so the chaplain has an accurate record to reflect upon when completing their 'chaplain final' questionnaire in relation to the relevant patient.

In week 7, the patient completes the 'Final' questionnaire and gives it to the champion. Independently, the chaplain also completes the chaplain's post intervention questionnaire, and gives it to the champion. The champion ensures all documents are securely stored and enters data into secure database online.

ANALYSIS The hypotheses will be tested in the following way.

Hypotheses

1. There will be a significant correlation between the number of times a chaplain sees a patient and the change in PROM scores from baseline to post intervention.

   Monotonicity will be checked using scatterplot and then parametric or non-parametric correlation will be used to test the relationship between the PROM scores and the number of times the patient has seen the chaplain. A significant correlation will show that there is a relationship between the number of chaplain visits and the change in the patient's self-reported outcomes between baseline and follow up.
2. There will be a significant correlation between the chaplain reported depth of the encounter and the change in PROM scores from baseline to post intervention.

   Monotonicity will be checked using scatterplot and then parametric or non-parametric correlation will be used to test the relationship between the PROM scores and the chaplain reported depth of the chaplaincy intervention. A significant correlation will show that there is a relationship between the chaplain's assessment of the depth of the intervention and the change in the patient's self-reported outcomes between baseline and follow up.
3. The patient experience of the chaplain encounter will be associated with the outcome of that intervention.

   Monotonicity will be checked using scatterplot and then parametric or non-parametric correlation will be used to test the relationship between the change in PROM scores and the self-reported quality of the chaplaincy intervention. A significant correlation will show that there is a relationship between the quality of the intervention and the self-reported outcomes.
4. There will be no difference in Scottish PROM scores according to whether patients self-describe as religious, spiritual, both, or neither

Two categories will be constructed. One will consist of all people who describe themselves as religious, spiritual or both. The second category will consist of those people who describe themselves as neither spiritual or religious. Independent samples t-tests will be used to determine whether changes in Scottish PROM scores are different according to whether people described themselves as religious/spiritual or not. One way ANOVA can also be used if samples are sufficient in all four groups.

Note, if there are multiple correlations and sufficient sample, a regression model can be constructed to develop predictors of positive chaplain interventions. The EQ5D data will be used where significant in constructing any multiple regression models.

Sample size calculation:

The effect size of chaplaincy intervention in palliative day care is difficult to estimate because there is no literature specific to this intervention. There are many anecdotal reports it has been very effective, and there is relevant comparable literature. For example there is evidence that spiritual interventions have 'significant moderate effect' in two separate recent meta-syntheses of the literature. 'Moderate' equates to a value of 0.3 to 0.5 using Cohen's d.

So, focusing on the primary hypotheses, allowing for testing twice on the same sample (Bonferroni correction: alpha = 0.025) with effect size 0.3, power 95%, G*Power version 2 calculated a necessary sample size of 156 in total.

ELIGIBILITY:
Inclusion Criteria:

* Patient attending the day unit for minimum 8 weeks
* Aged 18 and over

Exclusion Criteria:

* Patient unable to consent.
* Under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People referred to day care at participating hospices. All will be invited to participate excepting criteria above
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-01-18 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Scottish PROM | baseline to follow-up = 8 weeks
  The Scottish Patient Reported Outcome Measure is a five-item patient reported outcome measure of spiritual wellbeing. It generates a single score, minimum zero, maximum 20, representing spiritual wellbeing. The measure was validated to measure the impact of chaplain interventions. In a study of over 600 people who had seen a chaplain, scores ranged from 3 to 19, the mean was 12 and standard deviation 2.2. More work is required to calibrate the scale, but early indicators are positive in that scores appear normally distributed and the scale does not have ceiling or floor effects.

SECONDARY OUTCOMES:
EQ5D-3L | baseline to follow-up = 8 weeks
  Health related quality of life measure used around the world to estimate quality adjusted life years (QALYs). Here it is being used as a proxy measure of self reported health, because we do not have access to medical records and we may need a vicarious measure of wellness to factor in when analysing the results. It measures five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. The respondents self-rate their level of severity for each dimension using three levels (this is what the '3L' stands for)..

OTHER OUTCOMES:
'Depth' of chaplain encounter as recorded by chaplain | every week for 8 weeks
  Five point scale designed to indicate strength of connection between patient and chaplain. Devised by LOROS hospice, one represents the briefest of encounter to five representing support and prayer at death, to both patient and relatives. In more detail:
  One:
  Basic introduction/casual/ice breaker Two Talking about feelings and emotions Three Talking about the meaning of life, touching the spirituality of the patient Four Addressing spiritual need, eg., Praying, Holy Communion, connecting patient with faith communities.
  Five In depth spiritual care, eg.,end of life care, talking about death and dying, performing rituals.
  The scale has only been used in one hospice to date, and this study will further examine how it performs in practice.
Experience of chaplain encounter(s) as recalled by patient | At week 8 for each participant
  Four-item likert questions about 'what it was like' to be with the chaplain. These questions are not summated to form a scale, but are instead used to examine what part of the chaplain encounter appears to be most important to patients. These are the four items following the stem 'during my meeting with the chaplain I felt':
  1. I was listened to
  2. I was able to talk about what was on my mind
  3. My situation was understood
  4. My faith/beliefs were valued For example, in a 2018 study it was found that 'being able to talk about what was on my mind' was the most important element from patient perspective. (Snowden et al, 2018)

CONTACTS AND LOCATIONS:
Overall Officials: Austyn Snowden, PhD, Principal Investigator — Edinburgh Napier University
Locations (1):
- Strathcarron Hospice, Denny, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised datasets will be made available in line with local data protection policies.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Supporting information available now.
Access Criteria: Please contact Dr Paula Stevenson at p.stevenson@napier.ac.uk
URL: https://my.napier.ac.uk/Student-Administration/Research-Ethics-and-Governance/Documents/COPresearchintegrity_2013.pdf

REFERENCES:
- [Background] Snowden, A., Lobb, E. A., Schmidt, S., Swing, A., McFarlane, C., & Logan, P. (2018). What's on your mind? The only necessary question in spiritual care. Journal of the Study of Spirituality, 8(1), in press. http://doi.org/https://doi.org/10.1080/20440243.2018.1431031

DOCUMENTS (1):
  • Informed Consent Form (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/26/NCT03746626/ICF_000.pdf